CLINICAL TRIAL: NCT02464319
Title: Safety and Efficiency Study of Low-dose IL-2 Treatment in Primary Sjögren's Syndrome
Brief Title: A Phase II Study With Low-dose Recombinant Human IL-2 for the Treatment of Primary Sjögren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Monash University (Other); Beijing ShuangLu Pharmaceutical Co., Ltd. (Other)
Responsible Party: Principal Investigator, Zhanguo Li, Chief of Department of Rheumatology and Immunology,Peking University People's Hospital, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: hrIL-2-SS1
Record Dates: First submitted 2015-05-30; First posted 2015-06-08 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Primary Sjögren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: hrIL-2 active (Active Comparator): Intervention：Add hrIL-2 according to the protocol to original treatment. HrIL-2 active: 1 million U doses of human recombinant interleukin-2 s.c. injection
  Interventions: Drug: hrIL-2 active
- Placebo Comparator: hrIL-2 placebo (Placebo Comparator): 1 million U doses of placebo s.c. injection
  Interventions: Drug: hrIL-2 placebo

INTERVENTIONS:
Drug: hrIL-2 active — 1 million U doses of human recombinant interleukin-2 s.c. injection active group: placebo group =1:1
  Other Names: Human recombinant IL-2
  Arms: Experimental: hrIL-2 active
Drug: hrIL-2 placebo — 1 million U doses of placebo s.c. injection active group: placebo group =1:1
  Other Names: placebo
  Arms: Placebo Comparator: hrIL-2 placebo

SUMMARY:
Primary Sjögren's Syndrome (pSS) is an autoimmune disorder characterized by keratoconjunctivitis sicca and xerostomia. In addition, various extraglandular manifestations may develop. Several immunomodulating agents have been attempted in the treatment of pSS without achieving satisfactory results. Currently, there is no approved systemic treatment for pSS. Dysfunction of regulatory T (Treg) cells has been detected in diverse autoimmune diseases, which can be promoted by interleukin-2 (IL-2). The investigators hypothesized that low-dose IL-2 could be a novel therapy in active pSS patients. This clinical study will test the efficacy and safety of low dose IL-2 treatment in pSS. The investigators perform a single-centre, double-blind pilot trial with hrIL-2 in pSS. The investigators evaluate the effectiveness and safeness of low-dose hrIL-2 for primary Sjögren's Syndrome by randomized controlled study (hrIL-2 (N = 30) versus placebo group (N = 30)).

DETAILED DESCRIPTION:
Each pSS patients (n=60) with Scores>=6 on ESSDAI received low-dose IL-2 or placebo (active group: placebo group =1:1, 1 million units every other day subcutaneously (HrIL-2 1X 106, ip, Qod) for a period of 14 days. After a 14-day rest, another cycle started) for 3 cycles. The end points were safety, clinical and immunologic response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a primary Sjögren´s Syndrome
* ESSDAI score ≥ 6
* Liver values above 1,5 ULN
* Stable low dose systemic use of Glucocorticoids（<=7.5mg） in the last 4 weeks before begin with Study medication

Exclusion Criteria:

* Secondary Sjögren's Syndrome
* Pre-treatment with Cyclosporine A
* Receiving cyclosphosphamide, corticosteroid bolus with dose over 1 mg/kg, rituximab, belimumab, other immunosuppressives
* Infection
* Neoplasia
* Relevant cardiac, pulmonary, neurologic or psychiatric disease
* Life-Vaccination within 4 weeks before begin with study medication
* Pregnant or breast-feeding
* Weight under 45kg or more than 80kg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Examination of the therapeutic effects (improvement in ESSDAI) of low dose IL-2 in patients with primary Sjögren's Syndrome | 24 weeks

SECONDARY OUTCOMES:
Immunological Responses | 0,12,24weeks
  Analysis regulatory CD4+ T (Treg) cells , interleukin 17 (IL-17)-producing helper T (Th17) cells and follicular helper T (Tfh) cells before and during IL-2 treatment. P values below 0.05 are considered statistically significant in this study

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, MD, PhD, Principal Investigator — Peking University Institute of Rheumatology and Immunology
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Feng R, Xiao X, Wang Y, Huang B, Chen J, Cheng G, Jin Y. Metabolic impact of low dose IL-2 therapy for primary Sjogren's Syndrome in a double-blind, randomized clinical trial. Clin Rheumatol. 2024 Dec;43(12):3789-3798. doi: 10.1007/s10067-024-07165-2. Epub 2024 Oct 31. PMID 39482484
- [Derived] He J, Chen J, Miao M, Zhang R, Cheng G, Wang Y, Feng R, Huang B, Luan H, Jia Y, Jin Y, Zhang X, Shao M, Wang Y, Zhang X, Li J, Zhao X, Wang H, Liu T, Xiao X, Zhang X, Su Y, Mu R, Ye H, Li R, Liu X, Liu Y, Li C, Liu H, Hu F, Guo J, Liu W, Zhang WB, Jacob A, Ambrus JL Jr, Ding C, Yu D, Sun X, Li Z. Efficacy and Safety of Low-Dose Interleukin 2 for Primary Sjogren Syndrome: A Randomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2241451. doi: 10.1001/jamanetworkopen.2022.41451. PMID 36355371